CLINICAL TRIAL: NCT04392375
Title: Nifedipine XL Versus Placebo for the Treatment of Preeclampsia With Severe Features During Induction of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019H0431
Record Dates: First submitted 2020-05-02; First posted 2020-05-18 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Preeclampsia Severe
Keywords: preeclampsia severe, Nifedipine 30MG, placebo controlled
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Intervention Model Description: Patients are enrolled and randomly selected to receive Nifedipine or placebo through delivery of her infant.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nifedipine 30MG (Active Comparator): Oral administration of 30mg Nifedipine XL q24 hours until delivery
  Interventions: Drug: Nifedipine 30 MG
- Placebo (Placebo Comparator): Matching placebo group q24hrs until delivery
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Nifedipine 30 MG — Nifedipine XL is a long-acting medication used to lower blood pressure. The investigators want to learn whether women who receive the study drug will experience fewer severe-range blood pressure readings, and therefore need fewer intravenous (IV) medications to safely lower blood pressure.
  Arms: Nifedipine 30MG
Drug: Placebos — At the time of enrollment, patients will be randomized to either the study drug (oral Nifedipine XL 30mg) or identical placebo.
  Arms: Placebo

SUMMARY:
This is a randomized double blind placebo controlled trial comparing Nifedipine 30mg XL to placebo in 110 patients after decision has been made to proceed with induction of labor for the diagnosis of preeclampsia with severe features.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled trial comparing Nifedipine 30mg XL to placebo in 110 patients after decision has been made to proceed with induction of labor for the diagnosis of preeclampsia with severe features.

After diagnosis of preeclampsia with severe features and decision made to proceed with induction of labor. Patients were approached about study and if consented then were then randomized to placebo or nifedipine 30XL daily until delivery occurred.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 with a viable single or twin intrauterine pregnancy between 22 0/7 and 41 6/7 weeks gestation based on the best obstetric estimate by The American College of Obstetricians and Gynecologists (ACOG) criteria.
* Diagnosis of preeclampsia with severe features with decision made to induce labor. The patient may or may not have already received acute treatment for severe blood pressures.

Exclusion Criteria:

* Known allergy or adverse reaction to Nifedipine or any medical condition where Nifedipine is contraindicated, such as galactose intolerance, severe gastrointestinal (GI) structure, and GI hypomotility disorder.
* Currently receiving Nifedipine XL as part of hypertension management prior to induction of labor
* Participation in another trial that affects the primary outcome without prior approval
* Physician/provider or patient refusal
* Participation in this trial in a prior pregnancy
* Triplet or higher order pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cleary EM, Racchi NW, Patton KG, Kudrimoti M, Costantine MM, Rood KM. Trial of Intrapartum Extended-Release Nifedipine to Prevent Severe Hypertension Among Pregnant Individuals With Preeclampsia With Severe Features. Hypertension. 2023 Feb;80(2):335-342. doi: 10.1161/HYPERTENSIONAHA.122.19751. Epub 2022 Oct 3. PMID 36189646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nifedipine 30MG | Placebo
Started | 55 | 55
Completed | 53 | 49
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifedipine 30MG | Placebo | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [25 to 33.5] | 31 [24.4 to 34] | 30 [24.7 to 33.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 102
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 32 | 41 | 73
  Non-Hispanic Black | 15 | 3 | 18
  Hispanic | 5 | 4 | 9
  Non-Hispanic Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 53 | 49 | 102
Pregnancy BMI [Median (Inter-Quartile Range); unit: kg/m 2] | 32.9 [28 to 37.9] | 32.0 [25 to 36.1] | 32.45 [26.5 to 37]
BMI at delivery [Median (Inter-Quartile Range); unit: kg/m 2] | 37.8 [31.1 to 41.8] | 37 [29.9 to 40.7] | 37.4 [30.5 to 41.3]
Nulliparous [Count of Participants; unit: Participants] | 34 | 36 | 70
Chronic Hypertension [Count of Participants; unit: Participants] | 13 | 14 | 27
Chronic hypertension on maintenance medication (beta-blocker) [Count of Participants; unit: Participants] | 7 | 6 | 13
Smoking during current pregnancy [Count of Participants; unit: Participants] | 2 | 2 | 4
Diabates [Count of Participants; unit: Participants] | 12 | 8 | 20
Gestational age at delivery (week) [Count of Participants; unit: Participants]
  < 34 0/7 | 2 | 3 | 5
  34 0/7 - 36 6/7 | 28 | 25 | 53
  > 37 0/7 | 23 | 21 | 44
Neuraxial anesthesia [Count of Participants; unit: Participants] | 46 | 47 | 93
Twin gestation [Count of Participants; unit: Participants] | 2 | 2 | 4
Fetal Growth Restriction [Count of Participants; unit: Participants] | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Change in Blood Pressure (Both Systolic and Diastolic) Under the Treatment of NIfedipine 30mg XL Versus Placebo
Description: Measured acute antihypertension therapy between enrollment and delivery
Time Frame: Between enrollment and delivery, assessed up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine 30MG | Placebo
Number analyzed (Participants) | 53 | 49
Participants | 18 | 27

2. Secondary Outcome: Number of Participants Stratified by Route of Delivery
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine 30MG | Placebo
Number analyzed (Participants) | 53 | 49
Participants
  Cesarean Delivery | 11 | 17
  Vaginal Delivery | 42 | 32

3. Secondary Outcome: Number of Participants With Various Indications for Cesarean Delivery
Description: Some participants could have more than one indication for Cesarean Delivery.
Time Frame: Between enrollment and delivery, assessed up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine 30MG | Placebo
Number analyzed (Participants) | 11 | 17
Participants
  First stage arrest | 8 | 6
  Second stage arrest | 1 | 5
  Nonreassuring fetal status | 3 | 7
  Worsening maternal status | 2 | 1

4. Secondary Outcome: Number of Participants With Hypotension of ≥30% Decrease in Blood Pressure From Baseline Following Acute Antihypertensive Therapy
Time Frame: Between enrollment and delivery, assessed up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine 30MG | Placebo
Number analyzed (Participants) | 18 | 27
Participants | 8 | 6

5. Secondary Outcome: Number of Participants Who Required Acute Antihypertension Treatments Postpartum
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine 30MG | Placebo
Number analyzed (Participants) | 53 | 49
Participants | 20 | 19

ADVERSE EVENTS:
Time Frame: Between enrollment and delivery, assessed up to 18 weeks
Description: An adverse event (AE) will be defined as any untoward or unfavorable medical occurrence in a study participant, whether or not considered related to the subject's participation in the research.
Arm/Group | Nifedipine 30MG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04392375/Prot_SAP_000.pdf